CLINICAL TRIAL: NCT07103694
Title: Italian Real-life Multicenter Observational Study on Efficacy, Tolerability, and Safety of Innovative Drugs (Monoclonal Antibodies, Gepants, Ditans, Sumatriptan-naproxen) for Preventive or Acute Migraine Treatment.
Brief Title: i-NEED: NEw migrainE Drugs Database
Acronym: i-NEED
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 22/02
Record Dates: First submitted 2025-04-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Episodic Migraine; Chronic Migraine; Medication Overuse Headache
Keywords: migraine, anti-CGRP monoclonal antobodies, gepants, ditans, sumatriptan and naproxen combination
MeSH Terms: conditions — Headache Disorders, Secondary; Migraine Disorders | interventions — Calcitonin Gene-Related Peptide Receptor Antagonists; Naproxen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- individuals affected by migraine: episodic and chronic migraine
  Interventions: Drug: anti-CGRP monoclonal antibodies; Drug: gepants; Drug: combination of sumatriptan and naproxen; Drug: ditan

INTERVENTIONS:
Drug: anti-CGRP monoclonal antibodies — erenumab, fremanezumab, galcanezumab, eptinezumab
Drug: gepants — atogepant, rimegepant
Drug: combination of sumatriptan and naproxen — combination of sumatriptan and naproxen
Drug: ditan — lasmiditan

SUMMARY:
Approved by the Food and Drug Administration (FDA) and the European Medicine Agency (EMA) starting in 2018, anti-CGRP monoclonal antibodies (anti-CGRP mAbs) represent the first true revolution in the preventive treatment of migraine due to their selectivity and specificity. To date, four anti-CGRP mAbs have been developed for the preventive treatment of migraine: eptinezumab, erenumab, fremanezumab, and galcanezumab.Anti-CGRP mAbs constitute not only the first specific and selective treatment for the prevention of migraine but also the most extensively studied pharmacological category in this field, considering the vast and complex populations examined. The clinical effects of the various mAbs are substantially comparable and are characterized by several fundamental aspects:

* High efficacy in both episodic and chronic migraine, with the presence of super-responders who experience a reduction in the average monthly number of migraine days of >75% (or even 100%) compared to before treatment.
* Efficacy that is independent of the clinical form of migraine - with or without aura - and regardless of whether there is analgesic overuse.
* Efficacy maintained even in the presence of depressive or anxious comorbidities.
* Rapid onset of action (even more pronounced with eptinezumab), with the therapeutic effect appearing within the first week in most cases.
* Excellent tolerability with an absence of class-specific adverse events.
* Outstanding treatment adherence and a very low rate of treatment discontinuation in the long term. It should also be noted that the development of anti-drug antibodies or neutralizing antibodies to anti-CGRP mAbs is rare and does not significantly impact the efficacy or tolerability of treatment. Future clinical practice will need to clarify several additional aspects, such as: 1) whether treatment with anti-CGRP mAbs can modify the course of migraine; 2) the appropriate approach regarding any traditional preventive treatment (whether to continue or discontinue it); 3) the definition of the characteristics of non-responders; 4) the definition of patients with a delayed response to treatment.

Gepants are oral antagonists of the CGRP receptor. Among the four gepants synthesized so far (atogepant, rimegepant, ubrogepant, zavegepant), atogepant and rimegepant are currently available in Italy. Atogepant has proven to be an effective and well-tolerated option for the prevention of episodic and chronic migraines. Rimegepant is effective for both acute treatment and prevention of migraines, with a favorable safety profile and flexible oral administration. Lasmiditan is the first ditan effective for migraine attack and it represents a new therapeutic option for patients with contraindications to triptans, due to the presence of vascular risk factors, or for patients who experience undesirable side effects with these, thus increasing the therapeutic possibilities for the symptomatic treatment of migraine. The combination of sumatriptan 85 mg and naproxen sodium 500 mg is indicated for the acute treatment of migraine attacks in adult patients for whom sumatriptan monotherapy is insufficient.

DETAILED DESCRIPTION:
The European Headache Federation has published detailed guidelines on the state of the art regarding evidence of effectiveness in reducing the frequency and intensity of headache episodes, as well as the safety and tolerability of the four monoclonal antibodies under "ideal" experimental conditions, with patients selected based on stringent inclusion and exclusion criteria. This selection limits the direct transferability of the conclusions of these studies to clinical reality. Therefore, this study aims to evaluate, in a clinical practice setting, the real effectiveness in reducing the monthly frequency of migraine days and the tolerability and efficacy of monoclonal antibodies in a real-world evidence context. The study may later include all drugs that become available for this condition, subject to authorization by the competent Italian authority.

The present extension of the I-NEED study aims to integrate the collection and evaluation of real-life data on anti-CGRP monoclonal antibodies for migraine prophylaxis with the study of efficacy, safety, and tolerability-also in a real-world evidence context-of gepants in the prophylaxis of episodic and chronic migraine, and of rimegepant, ditans, and the sumatriptan-naproxen combination in the acute treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age more or equal 18 years;
* Males and females;
* Willingness to sign the informed consent;
* Episodic migraine for the use of drug indicated for migraine attack
* High frequency episodic migraine, at least 8 days per month of disabling migraine in the past 3 months;
* Chronic migraine, according to the ICHD-III criteria;

Exclusion Criteria:

* Other headaches different than migraine;
* Known intolerance to the eccipients;
* Vascular disease or Raynaud.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients include
  * adults (equal or more 18 years)
  * episodic or chronic migraine diagnosis,
  * treated with preventive or acute treatment drugs
Sampling Method: Non-Probability Sample
Enrollment: 2641 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
effectiveness of innovative drugs as migraine prophylaxis | the assessment will be conducted at 4 weeks from treatment initiation
  reduction in the number of monthly migraine days compared to the baseline average recorded in the three months preceding treatment
effectiveness of innovative drugs as migraine prophylaxis | the assessment will be conducted at 8 weeks from treatment initiation
  reduction in the number of monthly migraine days compared to the baseline average recorded in the three months preceding treatment
effectiveness of innovative drug as migraine prophylaxis | the assessment will be conducted at 12 weeks from treatment initiation
  reduction in the number of monthly migraine days compared to the baseline average recorded in the three months preceding treatment
effectiveness of innovative drugs as migraine prophylaxis | the assessment will be conducted at 24 weeks from treatment initiation
  reduction in the number of monthly migraine days compared to the baseline average recorded in the three months preceding treatment
effectiveness of innovative drugs as migraine prophylaxis | the assessment will be conducted at 48 weeks from treatment initiation
  reduction in the number of monthly migraine days compared to the baseline average recorded in the three months preceding treatment
2 hour-pain freedom | 2 hours
  Percentage of patients reporting complete pain relief within 2 hours after taking the innovative drug for migraine attack

SECONDARY OUTCOMES:
safety and tolerability of innovative drugs as migraine prophylaxis | the assessment will be conducted at 48 weeks from treatment initiation
  type and number of adverse events occurring during the study period (event details, duration, severity and action taken)
impact of innovative drugs as migraine prophylaxis on symptomatic medication use and medication overuse headache | the assessment will be conducted at 48 weeks from treatment initiation
  reduction in the average monthly consumption of analgesics in patients undergoing treatment with innovative drugs
impact of innovative drugs as migraine prophylaxis on migraine symptoms | the assessment will be conducted at 4 weeks from treatment initiation
  mean change in perceived pain intensity during a migraine attack (measured using the Numerical Rating Scale, score range 0-10) compared to the pre-treatment period
impact of innovative drugs as migraine prophylaxis on migraine symptoms | the assessment will be conducted at 8 weeks from treatment initiation
  mean change in perceived pain intensity during a migraine attack (measured using the Numerical Rating Scale, score range 0-10) compared to the pre-treatment period
impact of innovative drugs as migraine prophylaxis on migraine symptoms | the assessment will be conducted at 12 weeks from treatment initiation
  mean change in perceived pain intensity during a migraine attack (measured using the Numerical Rating Scale, score range 0-10) compared to the pre-treatment period
impact of innovative drugs as migraine prophylaxis on migraine symptoms | the assessment will be conducted at 24 weeks from treatment initiation
  mean change in perceived pain intensity during a migraine attack (measured using the Numerical Rating Scale, score range 0-10) compared to the pre-treatment period
impact of innovative drugs as migraine prophylaxis on migraine symptoms | the assessment will be conducted at 48 weeks from treatment initiation
  mean change in perceived pain intensity during a migraine attack (measured using the Numerical Rating Scale, score range 0-10) compared to the pre-treatment period
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 4 weeks from treatment initiation
  mean change in Headache Impact Test 6-TM scores (score range 36-78) before treatment
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 8 weeks from treatment initiation
  mean change in Headache Impact Test 6-TM scores (score range 36-78) before treatment
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 12 weeks from treatment initiation
  mean change in Headache Impact Test 6-TM scores (score range 36-78) before treatment
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 24 weeks from treatment initiation
  mean change in Headache Impact Test 6-TM scores (score range 36-78) before treatment
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 48 weeks from treatment initiation
  mean change in Headache Impact Test 6-TM scores (score range 36-78) before treatment
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 12 weeks from treatment initiation
  mean change in Migraine Disability Assessment Score Questionnaire (grade I: 0-5; grade II: 6-10; grade III: 11-20; grade IV>21) before treatment
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 24 weeks from treatment initiation
  mean change in Migraine Disability Assessment Score Questionnaire (grade I: 0-5; grade II: 6-10; grade III: 11-20; grade IV>21) before treatment
impact of innovative drugs as migraine prophylaxis on migraine-related disability | the assessment will be conducted at 48 weeks from treatment initiation
  mean change in Migraine Disability Assessment Score Questionnaire (grade I: 0-5; grade II: 6-10; grade III: 11-20; grade IV>21) before treatment
impact of innovative drugs as migraine prophylaxis on interictal disability | the assessment will be conducted at 4 weeks from treatment initiation
  Mean change in Migraine Interictal Burden Scale-4 (score range: 0-12)
impact of innovative drugs as migraine prophylaxis on interictal disability | the assessment will be conducted at 8 weeks from treatment initiation
  Mean change in Migraine Interictal Burden Scale-4 (score range: 0-12)
impact of innovative drugs as migraine prophylaxis on interictal disability | the assessment will be conducted at 12 weeks from treatment initiation
  Mean change in Migraine Interictal Burden Scale-4 (score range: 0-12)
impact of innovative drugs as migraine prophylaxis on interictal disability | the assessment will be conducted at 24 weeks from treatment initiation
  Mean change in Migraine Interictal Burden Scale-4 (score range: 0-12)
impact of innovative drugs as migraine prophylaxis on interictal disability | the assessment will be conducted at 48 weeks from treatment initiation
  mean change in Migraine Interictal Burden Scale-4 score (score range: 0-12)
impact of innovative drugs as migraine prophylaxis on work-related difficulties due to migraine | the assessment will be conducted at 12 weeks from treatment initiation
  mean change in the HEADWORK questionnaire score (two sections: the first one includes 13 items and the second one 12 items: every item requires a five point response scale ranging between 1-"no difficulty"-, 5 - "I cannot do it")
impact of innovative drugs as migraine prophylaxis on work-related difficulties due to migraine | the assessment will be conducted at 24 weeks from treatment initiation
  mean change in the HEADWORK questionnaire score (two sections: the first one includes 13 items and the second one 12 items: every item requires a five point response scale ranging between 1-"no difficulty"-, 5 - "I cannot do it")
impact of innovatine drugs as migraine prophylaxis on work-related difficulties due to migraine | the assessment will be conducted at 48 weeks from treatment initiation
  mean change in the HEADWORK questionnaire score (two sections: the first one includes 13 items and the second one 12 items: every item requires a five point response scale ranging between 1-"no difficulty"-, 5 - "I cannot do it")
impact of innovative drugs as migraine prophylaxis on economic resources in migraine | the assessment will be conducted at 12 weeks from treatment initiation
  mean change in the COSTI questionnaire score (evaluation of both direct and indirect cost directly gathered from patients)
impact of innovative drugs as migraine prophylaxis on economic resources in migraine | the assessment will be conducted at 24 weeks from treatment initiation
  mean change in the COSTI questionnaire score (evaluation of both direct and indirect cost directly gathered from patients)
impact of innovative drugs as migraine prophylaxis on economic resources in migraine | the assessment will be conducted at 48 weeks from treatment initiation
  mean change in the COSTI questionnaire score (evaluation of both direct and indirect cost directly gathered from patients)
patient subjective perception | the assessment will be conducted at 4 weeks from treatment initiation
  collection of subjective feedback from the patients regarding their experience with the medication, assessing patient satisfaction, ease of use of the medication perceived effectiveness with Patient Global Impression of Change (score range 1-7)
patient subjective perception | the assessment will be conducted at 8 weeks from treatment initiation
  collection of subjective feedback from the patients regarding their experience with the medication, assessing patient satisfaction, ease of use of the medication perceived effectiveness with Patient Global Impression of Change (score range 1-7)
patient subjective perception | the assessment will be conducted at 12 weeks from treatment initiation
  collection of subjective feedback from the patients regarding their experience with the medication, assessing patient satisfaction, ease of use of the medication perceived effectiveness with Patient Global Impression of Change (score range 1-7)
patient subjective perception | the assessment will be conducted at 24 weeks from treatment initiation
  assessment of subjective perception of change through Patient Global Impression of Change (score range 1-7)
patient subjective perception | the assessment will be conducted at 48 weeks from treatment initiation
  collection of subjective feedback from the patients regarding their experience with the medication, assessing patient satisfaction, ease of use of the medication perceived effectiveness with Patient Global Impression of Change (score range 1-7)
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 4 weeks from treatment initiation
  percentage of patients achieving a >50% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 8 weeks from treatment initiation
  percentage of patients achieving a >50% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 12 weeks from treatment initiation
  percentage of patients achieving a >50% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 24 weeks from treatment initiation
  percentage of patients achieving a >50% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 48 weeks from treatment initiation
  percentage of patients achieving a >50% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 4 weeks from treatment initiation
  percentage of patients achieving a >75% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 8 weeks from treatment initiation
  percentage of patients achieving a >75% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 12 weeks from treatment initiation
  percentage of patients achieving a >75% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 24 weeks from treatment initiation
  percentage of patients achieving a >75% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 48 weeks from treatment initiation
  percentage of patients achieving a >75% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 4 weeks from treatment initiation
  percentage of patients achieving a 100% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 8 weeks from treatment initiation
  percentage of patients achieving a 100% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 12 weeks from treatment initiation
  percentage of patients achieving a 100% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 24 weeks from treatment initiation
  percentage of patients achieving a 100% reduction in monthly migraine days compared to the pre-treatment period
response rates to innovative drugs as migraine prophylaxis | the assessment will be conducted at 48 weeks from treatment initiation
  percentage of patients achieving a 100% reduction in monthly migraine days compared to the pre-treatment period
1 hour-pain freedom | 1 hour after taking the innovative drug for migraine attack
  Percentage of patients reporting complete pain relief within 1 hour after taking the innovative drug for migraine attack
2 hours-pain relief | 2 hours after taking the innovative drug for migraine attack
  percentage of patients reporting a 50% reduction in pain intensity wiithin 2 hours after taking the innovative drug for migraine attack
disappearance of Most Bothersone Symptom | 2 hours after taking the innovative drug for migraine attack
  percentage of patients experiencing the disappearence of the Most Bothersone Symptom (the most disabling by the patient) within wiithin 2 hours after taking the innovative drug for migraine attack
presence or absence of associated symptoms (nausea, vomiting, photophobia, phonophobia) | 1-48 hours after taking the innovative drug for migraine attack
  presence or absence of associated symptoms (nausea, vomiting, photophobia, phonophobia) at predefined time intervals of 1, 2, 3, 4, 6, 8, 24 and 48 hours
24 hour-sustained pain freedom | 24 hours after taking the innovative drug for migraine attack
  percentage of patients experiencing complete pain relief within 2 hours after taking the innovative drug for migraine attack
24 hour-sustained pain relief | 24 hours after taking the innovative drug for migraine attack
  percentage of patients experiencing a 50% reduction in pain intensity within 2 hours after taking the innovative drug for migraine attack
headache recurrence | 2 hours after taking the innovative drug for migraine attack
  definition of the moment of possible migraine pain recurrence (headache recurernce), as well as its intensity within 24 and 48 hours following the administration of the medication (limited to patients who experienced pain freedom within 2 hours)
use of rescue medication | 24 hours after taking the innovative drug for migraine attack
  use of rescue medication and evaluation of the time interval between the first and the second dose
adverse occurence | 0-48 hours after taking the innovative drug for migraine attack
  definition of the type and number of adverse events occurring within 48 hours of taking the innovative drug for migraine attack (event details, duration, severity and action taken)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Rome, Italy, Italy

REFERENCES:
- [Background] Sacco S, Bendtsen L, Ashina M, Reuter U, Terwindt G, Mitsikostas DD, Martelletti P. European headache federation guideline on the use of monoclonal antibodies acting on the calcitonin gene related peptide or its receptor for migraine prevention. J Headache Pain. 2019 Jan 16;20(1):6. doi: 10.1186/s10194-018-0955-y. PMID 30651064
- [Background] Goadsby PJ, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Zhang F, Sapra S, Picard H, Mikol DD, Lenz RA. A Controlled Trial of Erenumab for Episodic Migraine. N Engl J Med. 2017 Nov 30;377(22):2123-2132. doi: 10.1056/NEJMoa1705848. PMID 29171821
- [Background] Reuter U, Goadsby PJ, Lanteri-Minet M, Wen S, Hours-Zesiger P, Ferrari MD, Klatt J. Efficacy and tolerability of erenumab in patients with episodic migraine in whom two-to-four previous preventive treatments were unsuccessful: a randomised, double-blind, placebo-controlled, phase 3b study. Lancet. 2018 Nov 24;392(10161):2280-2287. doi: 10.1016/S0140-6736(18)32534-0. Epub 2018 Oct 22. PMID 30360965
- [Background] Stauffer VL, Dodick DW, Zhang Q, Carter JN, Ailani J, Conley RR. Evaluation of Galcanezumab for the Prevention of Episodic Migraine: The EVOLVE-1 Randomized Clinical Trial. JAMA Neurol. 2018 Sep 1;75(9):1080-1088. doi: 10.1001/jamaneurol.2018.1212. PMID 29813147
- [Background] Detke HC, Goadsby PJ, Wang S, Friedman DI, Selzler KJ, Aurora SK. Galcanezumab in chronic migraine: The randomized, double-blind, placebo-controlled REGAIN study. Neurology. 2018 Dec 11;91(24):e2211-e2221. doi: 10.1212/WNL.0000000000006640. Epub 2018 Nov 16. PMID 30446596
- [Background] Dodick DW, Silberstein SD, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Effect of Fremanezumab Compared With Placebo for Prevention of Episodic Migraine: A Randomized Clinical Trial. JAMA. 2018 May 15;319(19):1999-2008. doi: 10.1001/jama.2018.4853. PMID 29800211
- [Background] Silberstein SD, Dodick DW, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Fremanezumab for the Preventive Treatment of Chronic Migraine. N Engl J Med. 2017 Nov 30;377(22):2113-2122. doi: 10.1056/NEJMoa1709038. PMID 29171818
- [Background] Dodick DW, Goadsby PJ, Silberstein SD, Lipton RB, Olesen J, Ashina M, Wilks K, Kudrow D, Kroll R, Kohrman B, Bargar R, Hirman J, Smith J; ALD403 study investigators. Safety and efficacy of ALD403, an antibody to calcitonin gene-related peptide, for the prevention of frequent episodic migraine: a randomised, double-blind, placebo-controlled, exploratory phase 2 trial. Lancet Neurol. 2014 Nov;13(11):1100-1107. doi: 10.1016/S1474-4422(14)70209-1. Epub 2014 Oct 5. PMID 25297013
- [Background] Lipton RB, Goadsby PJ, Smith J, Schaeffler BA, Biondi DM, Hirman J, Pederson S, Allan B, Cady R. Efficacy and safety of eptinezumab in patients with chronic migraine: PROMISE-2. Neurology. 2020 Mar 31;94(13):e1365-e1377. doi: 10.1212/WNL.0000000000009169. Epub 2020 Mar 24. PMID 32209650
- [Background] Lipton RB, Croop R, Stock EG, Stock DA, Morris BA, Frost M, Dubowchik GM, Conway CM, Coric V, Goadsby PJ. Rimegepant, an Oral Calcitonin Gene-Related Peptide Receptor Antagonist, for Migraine. N Engl J Med. 2019 Jul 11;381(2):142-149. doi: 10.1056/NEJMoa1811090. PMID 31291516
- [Background] Goadsby PJ, Wietecha LA, Dennehy EB, Kuca B, Case MG, Aurora SK, Gaul C. Phase 3 randomized, placebo-controlled, double-blind study of lasmiditan for acute treatment of migraine. Brain. 2019 Jul 1;142(7):1894-1904. doi: 10.1093/brain/awz134. PMID 31132795
- [Background] Brandes JL, Kudrow D, Stark SR, O'Carroll CP, Adelman JU, O'Donnell FJ, Alexander WJ, Spruill SE, Barrett PS, Lener SE. Sumatriptan-naproxen for acute treatment of migraine: a randomized trial. JAMA. 2007 Apr 4;297(13):1443-54. doi: 10.1001/jama.297.13.1443. PMID 17405970